CLINICAL TRIAL: NCT06579573
Title: ONO-2017 Phase III Study A Multicenter, Open-label Study in Japanese Patients With Primary Generalized Tonic Clonic Seizures.
Brief Title: ONO-2017 Study Japanese Patients With Primary Generalized Tonic Clonic Seizures.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONO-2017-01; jRCT2031210624 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2024-08-08; First posted 2024-08-30 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Epilepsy, Generalized
MeSH Terms: conditions — Epilepsy, Generalized | interventions — Cenobamate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cenobamate (Experimental)
  Interventions: Drug: Cenobamate

INTERVENTIONS:
Drug: Cenobamate — Cenobamate will be orally administered once daily.

SUMMARY:
To investigate the efficacy and safety of ONO-2017 in combination with antiepileptics in Japanese epileptic patients with generalized tonic-clonic seizures.

ELIGIBILITY:
Inclusion Criteria:

1. Gender and age: Japanese patients, regardless of gender, aged 12 years or older at the time of informed consent.
2. Subject has a clinical diagnosis of Primary Generalized Tonic-Clonic (PGTC) seizures in the setting of idiopathic generalized epilepsy.
3. Subject experiences at least 5 Primary Generalized Tonic-Clonic (PGTC) seizures in 12 weeks.
4. Subject is currently receiving 1 to a maximum of 3 concomitant Antiepileptic Drugs(AEDs) with fixed dosing regimens

Exclusion Criteria:

1. Subject has a history of status epilepticus that required hospitalization within 15 months prior to enrollment.
2. Subject has seizure clusters where individual seizures cannot be counted orclassified.
3. History of non-epileptic or psychogenic seizures.
4. Subject has a concomitant diagnosis of Partial Onset Seizure(POS).
5. Subject has a history of any serious drug-induced hypersensitivity reaction (including but not limited to Stevens Johnson syndrome, toxic epidermal necrolysis, drug reaction with eosinophilia and systemic symptoms(DRESS), Drug-induced hypersensitivity syndrome(DIHS)) or any drug-related rash requiring hospitalization.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-07-12 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Percentage Change in generalized tonic-clonic (PGTC) seizure frequency per 28-Day Interval | 12 Weeks of the Maintenance Phase
  Convert the frequency of generalized tonic-clonic seizures (PGTC) in the Maintenance Phase and Pre-treatment Phase to a 28-day interval. Calculate the percentage change for these.

SECONDARY OUTCOMES:
Percentage Change in all generalized seizure frequency per 28-Day | 12 Weeks of the Maintenance Phase
  Convert the frequency of all generalized seizures in the Maintenance Phase and Pre-treatment Phase to a 28-day interval. Calculate the percentage change for these.
Percentage of Subjects with Reduction in Generalized Seizure Frequency per 28-Day Interval | 12 Weeks of the Maintenance Phase
  The percentage of subjects who have a 50%, 75%, 90%, and 100% reduction in all generalized seizure frequency per 28-day interval during the Maintenance Phase relative to the Pre-treatment Phase

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (25):
- Japan (25):
  - Aichi Medical University Hospital, Aichi
  - Hospital of the University of Occupational and Environmental Health, Japan, Fukuoka
  - Southern TOHOKU Research Institute for Neuroscience Southern TOHOKU Medical Clinic, Fukushima
  - Local Independent Administrative Corporation Hiroshima City Hospital Organization Hiroshima City Hiroshima Citizens Hospital, Hiroshima
  - Hokkaido University Hospital, Hokkaido
  - Itami City Hospital, Hyōgo
  - Tsuchiura Kyodo General Hospita, Ibaraki
  - University of Tsukuba Hospital, Ibaraki
  - Kagoshima University Hospital, Kagoshima
  - SHOWA University Fujigaoka Hospital, Kanagawa
  - Yokohama City University Hospital, Kanagawa
  - National Hospital Organization Nishiniigata Chuo Hospital, Niigata
  - Koide Clinic of Epilepsy and Neurological Disorders, Osaka
  - TMG Asaka Medical Center, Saitama
  - NHO Shizuoka Institute of Epilepsy and Neurological Disorder, Shizuoka
  - Jichi Medical University Hospital, Tochigi
  - Jikei University Hospital, Tokyo
  - Maynds Tower Mental Clinic, Tokyo
  - National Center of Neurology and Psychiatry, Tokyo
  - Nihonbashi Neuro Clinic, Tokyo
  - Shinjuku Neuro Clinic, Tokyo
  - Tokyo Women's Medical University, Adachi Medical Center, Tokyo
  - Yamaguchi Grand Medical Center, Yamaguchi
  - University of Yamanashi Hospital, Yamanashi
  - Yamanashi Prefectural Central Hospital, Yamanashi

IPD SHARING:
Plan to Share IPD: No